CLINICAL TRIAL: NCT05841316
Title: The ED95 Dose Determined by Classical Train-of-four Ratio of Sugammadex to Reverse Rocuronium-Induced Deep Neuromuscular Block Back to Shallow Neuromuscular Block
Brief Title: The ED95 Dose of Sugammadex to Reverse Rocuronium-Induced Deep Neuromuscular Block Back to Shallow Neuromuscular Block
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Menekse Ozcelik, Associate Professor, Ankara University
Other Study IDs: 95
Record Dates: First submitted 2023-04-22; First posted 2023-05-03 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Deep Neuromuscular Blockade; Anesthesia, General
Keywords: neuromuscular block; sugammadex; ED95; rocuronium
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sugammadex ED95%: Sugammadex 0.6 mg/kg will be given in the first patient. The primary outcome is the success of recovery from deep (PTC:1-3) to superficial neuromuscular block (TOFR: 0.4) in 5 minutes after the administration of sugammadex.
  In case of success, the next patient will be given the same or reduced dose of 0.2 mg/kg sugammadex according to the randomisation scheme.
  In case of failure, the next patient will be given an increased dose of 0.2 mg/kg sugammadex.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — During the surgery, the desired level of neuromuscular block will be deep and followed by post-tetanic-count (PTC) of 1 to 3 in every 5 minutes. 0.3-1mg/kg/h rocuronium will be infused to ensure PTC of 1 to 3.
  At the end of the surgery, 0,6 mg sugammadex will be given as a bolus in the first patient of the study. The duration between the completion of sugammadex injection and the first measurement of Train-of-four ratio (TOFR) of 0.4 will be recorded.
  If the TOFR is achieved to 0.4 after sugammadex bolus of 0,6 mg/kg in 5 minutes, the result of reversal will be evaluated as positive. The consecutive patient will be given the same or decreased dose of sugammadex by 0,2 mg/kg according to the randomisation scheme.
  If the patient fails to recover from deep neuromuscular block to superficial block in 5 minutes after a given dose of sugammadex, the consecutive patient will be administered increased dose of sugammadex by 0,2 mg/kg.

SUMMARY:
In the European Society of Anaesthesiology and Intensive Care (ESAIC) guideline on the use of neuromuscular blockers published in 2023, it was suggested that sugammadex could be used to reverse deep and moderate neuromuscular blockade, and that neostigmine could be used to reverse superficial neuromuscular block (expressed as Train-of-Four Ratio (TOFR) 0.4 and above) to TOFR 0.9. Therefore, it has been hypothesized that a transition from deep neuromuscular block to superficial neuromuscular block can be achieved with lower than standard dose of sugammadex, followed by usual dose of neostigmine which results complete neuromuscular recovery from superficial neuromuscular block.

This study is planned with 2 stages. In the first phase of the study, the main goal is to determine the dose of sugammadex that would reverse the rocuronium induced deep neuromuscular block (PTC 1 to 3) to superficial neuromuscular block (TOFR: 0.4) in 95% of patients in 5 minutes following administration.

DETAILED DESCRIPTION:
Laparoscopic surgery also known as minimally invasive surgery is a type of surgical procedure which allows a surgeon to access the inside of the abdomen and pelvis without having to make large incisions in the skin. As the administration of deep neuromuscular block has been shown to improve surgical conditions in laparoscopic abdominal surgery, patients are usually kept under deep neuromuscular block using either intermittent bolus or continous infusion of neuromuscular blocking drugs such as rocuronium during the surgical procedure (1). Due to small incisions of fascia and skin, the duration between the completion of intra-abdominal surgical manipulation in which the patient is usually under rocuronium-induced deep neuromuscular block (RIDeNB) and the end of skin sutures in which the patient should be closed to fully recover from RIDeNB is often short. However, the time interval required for reversing RIDeNB may be quite longer if spontaneous neuromuscular recovery is allowed. Therefore, sugammadex of 4 mg/kg is usually recommended to shorten the duration of RIDeNB reversal (2).

The incidence of an unplanned re-intubation which occurs shortly after a failed extubation is approximately 0.04-0.09% (3,4). Although the incidence seems quite low, it may be a life threatening adverse event. In case of unplanned re-intubation after the administration of 4 mg/kg sugammadex to reverse RIDeNB, the anesthesiologist may choose to give a non-steroidal neuromuscular blocker or 1,2 mg/kg of a high dose of rocuronium. With re-administration of 1.2 mg/kg rocuronium up to 30 minutes after sugammadex administration, the onset of neuromuscular blockade again may be prolonged to approximately 4 minutes and also the duration of neuromuscular blockade may be shortened to approximately 15 minutes. Due to the possibility of re-intubation after every single extubation, the lower the dose of sugammadex administered during the recovery phase of RIDeNM, the less the need for the dose of rocuronium to be applied for the next intubation attempt or better re-intubation conditions will be provided even if the same dose is applied. To lower the standard reversal dose of sugammadex, it is assumed that gradual recovery can be achieved with the combination of sugammadex and neostigmine to achieve a complete neuromuscular recovery with an effective, reliable and lower cost manner.

In the ESAIC guideline on the use of neuromuscular blockers published in 2023, it was suggested that sugammadex could be used to reverse deep and moderate neuromuscular blockade, and that neostigmine could be used to reverse superficial neuromuscular block (expressed as TOFR 0.4 and above) to TOFR 0.9 (5). Therefore, it has been hypothesized that a transition from deep neuromuscular block to superficial neuromuscular block can be achieved with lower than standard dose of sugammadex, followed by usual dose of neostigmine which results complete neuromuscular recovery from superficial neuromuscular block.

This study is planned with 2 stages. In the first phase of the study, the main goal is to determine the dose of sugammadex that would reverse the rocuronium induced deep neuromuscular block (PTC 1 to 3) to superficial neuromuscular block (TOFR: 0.4) in 95% of patients in 5 minutes following administration.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5-24.9 kg/m2
* ASA 1 and 2
* Patients undergoing elective surgery

Exclusion Criteria:

* Allergic reactions to study drugs
* Planned rapid sequence anesthesia induction
* Patient refusal
* Emergence surgery
* Neuromuscular diseases
* Renal disease or failure with elevated creatinine above 2.0 mg/dL
* Liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ASA 1 and 2 patients undergoing elective surgery with normal BMI
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
ED95 of sugammadex | 5 minutes
  The dose of sugammadex to provide reversal from deep to superficial rocuronium induced neuromuscular blockade in 5 minutes after bolus administration in 95% of patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fuchs-Buder T, Schmartz D, Baumann C, Hilt L, Nomine-Criqui C, Meistelman C, Brunaud L. Deep neuromuscular blockade improves surgical conditions during gastric bypass surgery for morbid obesity: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jul;36(7):486-493. doi: 10.1097/EJA.0000000000000996. PMID 30985536
- [Result] Chen S, Zhang Y, Che L, Shen L, Huang Y. Risk factors for unplanned reintubation caused by acute airway compromise after general anesthesia: a case-control study. BMC Anesthesiol. 2021 Jan 12;21(1):17. doi: 10.1186/s12871-021-01238-4. PMID 33435881
- [Result] Banik RK, Honeyfield K, Qureshi S, Reddy SG. Incidence and Mortality Rate of Perioperative Reintubation: Case Series of 196 Patients. AANA J. 2021 Dec;89(6):476-479. PMID 34809752
- [Result] Fuchs-Buder T, Romero CS, Lewald H, Lamperti M, Afshari A, Hristovska AM, Schmartz D, Hinkelbein J, Longrois D, Popp M, de Boer HD, Sorbello M, Jankovic R, Kranke P. Peri-operative management of neuromuscular blockade: A guideline from the European Society of Anaesthesiology and Intensive Care. Eur J Anaesthesiol. 2023 Feb 1;40(2):82-94. doi: 10.1097/EJA.0000000000001769. Epub 2022 Nov 15. PMID 36377554